CLINICAL TRIAL: NCT06844110
Title: Application of 68GA-labeled CD73 Targeting Probe PET/CT Imaging in the Diagnosis of Malignant Tumor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-CD73-2
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Tumor Immunity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malignant tumor (Experimental)
  Interventions: Drug: 68GA-DOTA-dPNE

INTERVENTIONS:
Drug: 68GA-DOTA-dPNE — Intravenous administration of 68GA-DOTA-dPNE tracer

SUMMARY:
68Ga-DOTA-dPNE PET/CT imaging was performed on patients with malignant tumors to observe the binding of lesions with the tracer and evaluate the expression of CD73. At the same time, correlation analysis was performed combined with relevant clinical indicators to evaluate the efficacy of 68Ga-DOTA-dPNE in the diagnosis and guidance of malignant tumor patients, and predict the response of targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age: ≥18 years, expected survival ≥12 weeks 2: Without radiotherapy and chemotherapy, surgery or biopsy is feasible to obtain pathological diagnosis 3: Standard Solid Tumor Response Evaluation Criteria (RECIST) version 1.1 with at least one measurable target lesion 4: Obtain written informed consent and be able to follow up

Exclusion Criteria:

- 1: Severe liver and kidney dysfunction. 2: Women who are planning to conceive, pregnant, or breastfeeding, as well as those planning to have children during the study period, are not eligible to participate in this research. Women of childbearing potential must use effective contraception throughout the course of the study.

3: Individuals unable to lie flat for thirty minutes. 4: Suffers from claustrophobia or other mental illnesses 5: Researchers believe that the subject has other conditions that make them unsuitable for inclusion in this study 6: Refuses to join this clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Lesion SUV value | After the completion of the PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Xianzhong Zhang, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- PUMCH, Dongcheng, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No